CLINICAL TRIAL: NCT01892332
Title: The Effective Concentration of Lidocaine With Fentanyl in Lumbar Epidural Anesthesia for Transurethral Resection of Prostate(TURP) in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2013-0257
Record Dates: First submitted 2013-06-30; First posted 2013-07-04 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: BPH( Benign Prostate Hyperplasia); TURP(Transurethral Resection of Prostate)
MeSH Terms: interventions — Anesthesia, Epidural; Lidocaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- lidocaine with fentanyl 75ug (Other)
  Interventions: Drug: epidural block with lidocaine and fentanyl

INTERVENTIONS:
Drug: epidural block with lidocaine and fentanyl — The study method was a step-up/step-down sequence model where the dose for following patients was determined by the outcome of the preceding block. The starting concentration of lidocaine was 1.5 % mixed with fentanyl 75 ug. All patients receive 13mL of lidocaine with fentanyl 75ug. The concentration of lidocaine for subsequent patients is determined by the outcome in the previous patient according to up and down sequential allocation in 0.1% increments. In the case of block failure, the concentration of lidocaine was increased by 0.1%.
  Conversely, block success resulted in a reduction in concentration by 0.1%.

SUMMARY:
Epidural lidocaine is widely used in anesthesia for urologic or lower abdominal surgery because of its rapid onset. But the epidural anesthesia using high concentration of lidocaine may cause excessive motor block and unwanted side effects such as nausea, vomiting and hypotension.

This is a study to determine the effective concentration of lidocaine with fentanyl in lumbar epidural anesthesia for transurethral resection of prostate in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 -3, patients scheduled for TURP( transurethral resection of prostate) were included

Exclusion Criteria:

* Patients with any contraindication to epidural anesthesia were excluded.

  * cognitive impairment
  * coagulopathy
  * allergy to lidocaine
  * infection at the puncture site

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Determining the effective concentration of lidocaine with fentanyl in lumbar epidural anesthesia for transurethral resection of prostate(TURP) in elderly patients | A blinded Assistant assess sensory and motor blockade in a 2-min intervals up to 60 minutes.
  The occurrence of sensory block up to at T 12 and motor function score of 3 or more on the modified Bromage scale were considered characteristics of a successful block. Moreover, the surgery should be concluded without any complementary analgesia to confirm the success of the anesthetic procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea